CLINICAL TRIAL: NCT02399098
Title: The Effectiveness of Attentional Strategies on Throwing Performance and Gaze Behavior of Self-paced Tasks Under Fatigue and Non-fatigue Conditions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Wingate Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 0016-15-HYMC
Record Dates: First submitted 2015-03-15; First posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Motor Learning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- External focus group (Experimental): This group will be given instructions on how to focus on the external cue relevant to the task (e.g., focus on the center of the dart board).
  Interventions: Behavioral: Attentional focus
- Internal focus group (Experimental): This group will be instructed how to focus on the arm movements (e.g., feel the bend in your elbow).
  Interventions: Behavioral: Attentional focus
- Control (No Intervention): This group will be given general instructions on throwing techniques (e.g., hold the dart with four fingers and make sure it is in a stable position) but no attentional focus instructions will be given.

INTERVENTIONS:
Behavioral: Attentional focus — The participants will learn the dart throwing task according to specific instructions. Participants in all groups will be given the same technical instructions on how to throw the dart. The technical instructions will be followed by attentional focus instructions that will differ between the groups.
  Arms: External focus group; Internal focus group

SUMMARY:
Focusing attention is pertinent to the performance of closed self-paced motor tasks. The following study will examine the effectiveness of internal and external focus of attention instructions on the performance of a dart throwing task under rested and fatigue (after performing intense exercise) conditions. As well as the relationship between attentional focus instructions and gaze behavior under these two conditions.

DETAILED DESCRIPTION:
The participants will arrive at the Ribstein Center for Sports Medicine and Research at the Wingate Institute on four different occasions, 2-3 days apart, in order to complete three motor learning phases. Session 1 and 2 will include the acquisition phase, Session 3 will include the retention and transfer phases, and the last visit, Session 4, will include the fatigued session.

Sessions 1 and 2 The participants will be informed of the purpose, methods, and study protocol. Then an informed consent form will be provided to the participant to be signed. The participants will learn the throwing task according to specific instructions. Participants in all groups will be given the same technical instructions on how to throw the dart. The technical instructions will be followed by attentional focus instructions that will differ between groups. After receiving the instructions, the participants in both these groups will be given a questionnaire to fill in. The researcher will go over the answers with each participant to ensure that the instructions were understood. If needed, the instructions will be repeated until appropriate understanding and performance is achieved. Then, a 3-min practice period will begin. The participants of the internal focus group will be asked to perform the throwing movement of the arms 20 times without holding the dart. The external focus group's participants will be asked to perform the throwing motion 20 times while holding the dart. The participants in the control group will be asked to practice their stance, posture, and the holding of the dart.

Testing will begin after the preparation period. The Mobile Eye gaze tracking system will be fitted and calibrated to six different reference locations. The calibration target will be a board with six "X" shapes spaced 30 cm apart on a white paper that will be placed on the target. The external video will be located perpendicular to the participant in a way that the upper body and the arm movement can be seen in the frame. The participant will then perform the dart throwing task of 5 blocks of 12 trials, with a 2-min rest in between each block of trials. During the 2-min rest interval the researcher will remind each participant to use the attenational focus strategy. During the rest interval between the blocks, the system's calibration will be checked and calibrated again if necessary. In total, each participant will complete 120 trials of the dart throwing task in the acquisition phase.

Session 3 Upon arrival to the Lab, participants will be fitted with the Mobile Eye system, and calibration will be performed. The external video camera will be turned on and the participants will perform the same dart throwing task for 2 blocks of 10 trials, with 2min of rest in between. A transfer task will be performed after a 15-min break. Participants will be re-fitted with the Mobile Eye and re-calibration will be performed. The transfer task (an underarm throw) will be performed for 2 blocks of 10 trials with 2-min of rest in between.

Session 4 On the fourth and final visit, the participants will be randomly assigned into two groups. Each subgroup will perform two blocks of 10 trials, with a 60-sec rest in between, under different types of anaerobic physical exertions: (1) Leg Anaerobic condition (WAnT-leg): using the modified WAnT, and (2) Arm anaerobic condition (WAnT-arm): using the WAnT arm modification.

Before commencing the exercise test protocol, anthropometric measures will be determined for each participant. Height and body mass will be measured using a stadiometer (Seca, Birmingham, UK) and a digital scale (Model HBF-514C, Omron Healthcare Inc, Bannockburn, Illinois), respectively, and will be recorded to the nearest 0.1 cm and 0.1 kg, respectively. Skinfold thickness will be measured in triplicate using Caliper (Skyndex System 1, Caldwell, Justiss & Company, Inc, Fayetteville, Arkansas, USA). The following sites will be evaluated: biceps, triceps, subscapular, and suprailiac. Adiposity (percentage of body fat) will be estimated from the appropriate skinfold measurements using Durning and Womersly equations (Durnin & Womersley, 1974). All measurements will be performed by the same investigator. Preceding the anthropometric measurement and before beginning either test, either ergometer will be individually adjusted to fit each participant's height and body size. A heart rate monitor (Polar FT1, Polar Electro, USA) will be worn by each subject in order to record heart rate data. The eye tracking system will be put on and calibrated. Then the participants will remove the apparatus and will begin the physical exertion test. Subsequently, the participants will warm up for the WAnT-leg (men=75 W; women=50 W) and for the WAnT-arm (men=30 W; women=unloaded) by exercising at 60 rpm for 5 min.

During the warm-up period, participants will be asked to perform three all-out 5-sec sprints on the command of the researcher. Following the warm-up, participants will rest quietly for 10 min. Then the participants will perform ten consecutive 10 seconds sprints interspersed with 15 seconds recovery intervals. The participant will be instructed to sprint as fast as possible for 10 seconds. Verbal encouragement will be given during the test. The resistance for men will be set at 0.931 and 0.601 N/Kg-1, and for women 0.833 and 0.470 N/Kg-1 during the WAnT-leg and the WAnT-arm, respectively (Weber, Chia, & Inbar, 2006). Participants will be instructed to remain seated throughout the test and will be given verbal encouragement to maintain an all-out effort throughout the 10 seconds sprints. During each sprint, peak and mean power outputs will be calculated. Peak power (PP) will be the highest power produced in a 1 sec segment of each 10 seconds sprint, whereas mean power (MP) will be calculated as the average power during the 10 seconds duration. PP and MP will be expressed in watts and relative to body mass (W/Kg). A fatigue index (FI) will be calculated as the absolute difference between the PP and the MP divided by the PP and expressed in percentage (%FI). In order to monitor the exercise intensity during each exertion protocol, the following measures will be obtained prior to the beginning of the test, at the end of the last 10 seconds sprint and 3min and 5min after the last sprint: heart rate, lactate levels, and rate of perceived exertion. Five minutes after completing the WAnT-leg or-arm test, the participants will put on the eye tracking apparatus; if needed the system will be re-calibrated. Then the subject will be asked to perform the throwing task without additional explanation. This time period was chosen based on previous studies that found peak lactate after the WAnT test to occur following approximately 5 min of recovery (Weinstein, Bediz, Dotan, & Falk, 1998). At the end of the fourth session, participants will be asked to fill in the learning strategies' implementation questionnaire. This 4-questions questionnaire will include two close-ended questions and two open-ended questions, and is meant to check whether participants used their assigned attentional focus strategies.

ELIGIBILITY:
Inclusion Criteria:

* Participation in physical activity up to three hours per week presently and in the previous year.
* No previous experience in dart throwing

Exclusion Criteria:

* Attention deficit disorder
* Muscular function disorder
* Chronic/frequent use of medications that could affect neuromuscular function
* Injury to the dominant hand
* Being either elite athlete or sedentary

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Absolute error | Two weeks
  A measure of overall accuracy in performance - the distance from the target for each shot, without regard to direction
Variable error | Two weeks
  Performance variability - the standard deviations of the cluster of target hits
Quiet eye duration | Two weeks
  The length of time in milliseconds in which the performer's gaze is stable on the target

SECONDARY OUTCOMES:
Number of saccades | Two weeks
Number of fixations | Two weeks
Attentional focus comprehension | Two weeks
  A questionnaire will be given in order to assess the participants' understating and implementation of the instructions given.

CONTACTS AND LOCATIONS:
Overall Officials: Eias Kassem, MD, Principal Investigator — Hillel Yaffe Medical Center